CLINICAL TRIAL: NCT03355404
Title: Evaluate the Impact of the "Standing Patient" Pathway on Preoperative Anxiety.
Brief Title: Impact of the "Standing Patient" Pathway on Preoperative Anxiety.
Acronym: ANXIPADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A01253-50
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Standing Patient" (Experimental)
  Interventions: Other: standing patient
- "Standardized management in stretcher" (No Intervention)

INTERVENTIONS:
Other: standing patient — patient goes standing to the surgery room
  Arms: "Standing Patient"

SUMMARY:
For 25 years, the concept of Rapid Rehabilitation After Surgery or RRAC has developed to bring about a global care of the patient by establishing a safe and quality climate. With this concept of RRAC or fast track surgery, it is the idea that a patient will recover sooner than he is lying later. "Fast care" is based on the principle that any patient is valid before he / be operated and therefore do not need to come to a bed in the operating room.

The ambulatory surgery department of the CHU of Caen welcomes and supports adults and children over 8 years old. The following specialties are covered: dental surgery and stomatology, digestive and visceral surgery, orthopedic surgery, otolaryngological surgery, vascular surgery, gynecological surgery, urological surgery. The ambulatory surgery unit is experimenting with patient support at the operating theater on foot by the service stretcher team since December 2015. It seems that this technique makes it possible to improve the quality of care by respecting the dignity and autonomy; in fact to wander the patient preserves his glasses, his hearing aids, capillary prosthesis ... The patient is an actor and not dependent, he is accompanied and not taken away. The preservation of autonomy improves their feelings, especially in terms of dignity. It also appears to be a technique for participating in the reduction of preoperative anxiety, an important factor for postoperative follow-up.

However, studies reporting the benefit of this technique have rather evaluated the feelings of patients. To the best of our knowledge, there are no studies that have evaluated their benefit on anxiety reduction by questionnaires or ad hoc scales. Assessing anxiety with appropriate tools seems essential to determine a real impact.

We hypothesize that accompanying the patient to the operating room on foot would reduce preoperative anxiety. We have not yet found any studies showing that the "standing patient" pathway had an impact on preoperative anxiety. We propose to carry out a randomized study comparing the anxiety score using the APAIS scale at the operating room installation between patients benefiting from the "standing patient pathway" versus the patients receiving the care standard, that is to say the stretcher transport to the operating theater.

The duration of this study is evaluated at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Major patient.
* Patient hospitalized for surgery.
* Patient supported in the south block.
* Patients agreeing to participate in the study.
* Patient speaking and understanding French.

Exclusion Criteria:

* Patient with reduced mobility.
* Patient with a mental disability.
* Patient suffering from a severe psychiatric pathology.
* Major patient protected.
* Patient does not speak or understand French.
* Refusal of the patient to participate in the study.
* Patient who has been premedicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
APAIS score to the operating room installation | baseline
  APAIS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No